CLINICAL TRIAL: NCT00539279
Title: Treatment of Older Veterans With Chronic Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDA-2-009-07S
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Combat Disorders; Post-traumatic Stress Disorder
Keywords: Cognitive- Behavior Therapy; Combat Disorders; Elderly; Geriatrics; Implosive therapy; Neuropsychological Test; Post-traumatic Stress Disorder; Psychotherapy; Randomized Controlled Trial; Relaxation techniques
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic | interventions — Implosive Therapy; Floods; Relaxation Therapy; Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Exposure Therapy (PE) (Experimental): Prolonged Exposure Therapy (PE)
  Interventions: Behavioral: Prolonged Exposure Therapy (PE)
- Relaxation Training (RT) (Active Comparator): Relaxation Training (RT)
  Interventions: Behavioral: Relaxation Training (RT)

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy (PE) — PE is a therapy that aims to reduce PTSD symptoms via a systematic exposure to feared memories (by imaginal exposure - repeated narration about the traumatic memory) and situations (by in vivo exposure - engaging in feared but safe activities or facing feared situations).
  Other Names: Implosive therapy; flooding; systematic desensitization
  Arms: Prolonged Exposure Therapy (PE)
Behavioral: Relaxation Training (RT) — RT aims to teach relaxation methods in an effort to reduce anxiety. RT includes Progressive Muscle Relaxation, Imagery Rehearsal, and breathing training.
  Other Names: Progressive Muscle Relaxation; Breathing training
  Arms: Relaxation Training (RT)

SUMMARY:
This project represents the first randomized clinical trial of psychotherapy for older veterans with posttraumatic stress disorder (PTSD). It will compare relaxation training (RT) to prolonged exposure therapy (PE). The project will also examine whether cognitive impairment influences psychotherapy outcome.

Primary hypotheses: (1) Subjects in the PE condition will have significantly less severe PTSD symptoms, depressive symptoms, and functional impairment than subjects in the RT condition at posttest; (2) Executive functioning will modify the response to both treatments, such that those with impaired executive functioning will demonstrate a smaller reduction in PTSD symptoms (representing less clinically significant change).

DETAILED DESCRIPTION:
PTSD is associated with high rates of mortality from suicide and health complications, high healthcare costs, and diminished health and quality of life. Many military veterans have PTSD due to combat, and many veterans continue to carry the symptoms of PTSD into late life. The percentage of older veterans is expected to increase substantially in coming years (especially as Vietnam-era veterans become older adults). The psychosocial intervention with the most rigorous empirical support for treating PTSD in the general population is a cognitive-behavioral treatment known as exposure therapy (which involves helping patients face feared memories and situations), yet there have been no controlled studies of any psychosocial interventions for PTSD in samples of older adults. Some have argued that older adults will not respond well to exposure because of their cognitive limitations. However, several empirical studies have shown exposure therapy to be safe and effective with older adults with anxiety disorders other than PTSD.

The current project represents the first randomized clinical trial of psychotherapy for older veterans with posttraumatic stress disorder (PTSD). It will compare relaxation training (RT) to prolonged exposure therapy (PE). The project will also examine whether cognitive impairment influences psychotherapy outcome. The five-year Research Plan is divided into three phases. Phase 1 (Year 1) involves the development of procedures for assessment and preparation for the clinical trial. Phase 2 (Years 2-4) will entail the first randomized clinical trial of psychosocial treatments for PTSD in late life. One hundred veterans aged 60 years or older, with chronic PTSD, will be recruited from the San Diego VA PTSD Clinical Team and randomly assigned to 12 sessions of PE or 12 sessions of RT. Phase 3 (Year 5) will be comprised of final data collection, scoring and interpretation of all neuropsychological tests, data cleaning and analysis, and writing for publication of results. Primary hypotheses: (1) Subjects in the PE condition will have significantly less severe PTSD symptoms, depressive symptoms, and functional impairment than subjects in the RT condition at posttest; (2) Executive functioning will modify the response to both treatments, such that those with impaired executive functioning will demonstrate a smaller reduction in PTSD symptoms (representing less clinically significant change).

ELIGIBILITY:
Inclusion Criteria:

* Veterans with primary diagnosis of chronic PTSD due to combat or non-sexual military trauma; comorbid mood and anxiety disorders are expected, and will be permitted (to maximize generalizability) if PTSD symptoms are judged to be predominant based on primacy and severity of symptoms
* Male
* Age 60 or older; and
* English literacy.

Exclusion Criteria:

* Unmanaged psychosis or manic episodes in past year
* Substance dependence or alcohol dependence in past 3 months
* Concurrent psychotherapies targeting PTSD or exposure therapy for other anxiety symptoms [veterans who are engaged in treatment for non-PTSD symptoms (e.g., 12-step programs for substance problems) will be eligible]
* Severe cardiovascular or respiratory disease that would make it difficult to ensure regular attendance at psychotherapy sessions
* Probable dementia (based on chart diagnosis); or
* Head trauma resulting in loss of consciousness longer than 20 minutes.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Thorp, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Walter KH, Glassman LH, Wells SY, Thorp SR, Morland LA. The Impact of Depression Severity on Treatment Outcomes Among Older Male Combat Veterans with Posttraumatic Stress Disorder. J Trauma Stress. 2020 Jun;33(3):345-352. doi: 10.1002/jts.22503. Epub 2020 Mar 26. PMID 32216149
- [Derived] Thorp SR, Glassman LH, Wells SY, Walter KH, Gebhardt H, Twamley E, Golshan S, Pittman J, Penski K, Allard C, Morland LA, Wetherell J. A randomized controlled trial of prolonged exposure therapy versus relaxation training for older veterans with military-related PTSD. J Anxiety Disord. 2019 May;64:45-54. doi: 10.1016/j.janxdis.2019.02.003. Epub 2019 Feb 21. PMID 30978622
- See also: Click here for more information about this study: Treatment of Older Veterans with Chronic Posttraumatic Stress Disorder — http://ptsdstudies.weebly.com/study-3-older-adults.html

RESULTS

PARTICIPANT FLOW:
Period: Treatment
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT)
Started | 41 | 46
Completed | 30 | 38
Not Completed | 11 | 8
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Death | 1 | 0
Period: Post-Treatment Assessment
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT)
Started | 30 (Individuals eligible for post-treatment assessment (includes all individuals randomized to PE)) | 38 (Individuals eligible for post-treatment assessment (includes all individuals randomized to RT))
Completed | 18 | 29
Not Completed | 12 | 9
Not completed — Lost to Follow-up | 12 | 9
Period: 6-Month Follow-Up Assessment
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT)
Started | 18 (Individuals eligible for 6-month assessment (includes all individuals randomized to PE)) | 29 (Individuals eligible for 6-month assessment (includes all individuals randomized to RT))
Completed | 17 | 22
Not Completed | 1 | 7
Not completed — Lost to Follow-up | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT) | Total
Number analyzed (Participants) | 41 | 46 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.51 (6.21) | 64.44 (4.49) | 65.54 (5.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 41 | 46 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 39 | 41 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 31 | 38 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 41 | 46 | 87
PTSD Checklist (PCL) [Mean (Standard Deviation); unit: units on a scale] — The PTSD Checklist is a self-report questionnaire about PTSD symptoms. The version used in this study is called the PCL-S, which denotes a specific traumatic event for subjects to respond to. There are 17 items, each with response categories from 1 to 5. Thus, the total score ranges from 17 to 85. Higher scores reflect higher levels of PTSD symptoms, and a score of 50 or above is commonly interpreted to designate clinically significant PTSD symptoms.
  units on a scale | 57.46 (12.66) | 59.98 (11.80) | 58.28 (12.36)
Patient Health Questionnaire Depression Subscale (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 is a self-report questionnaire about depressive symptoms. There are 9 scored items, each with response categories from 0 (zero) to 3. Thus, the total score ranges from 0 to 27. Higher scores reflect higher levels of depressive symptoms, with interpretation as follows:
  0 (zero) No depression 1-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression
  units on a scale | 12.13 (6.57) | 15.12 (5.17) | 13.28 (6.20)
Clinician-Administered PTSD Scale Severity Score (CAPS) [Mean (Standard Deviation); unit: units on a scale] — The CAPS is a clinician-administered interview about PTSD symptoms. There are 17 scored items for PTSD severity, each with response categories from 0 (zero) to 4 separately for both frequency and severity. Thus, each item can receive a score of 0 (zero) to 8, and the total severity score ranges from 0 to 136. Higher scores reflect higher levels of PTSD symptoms. Scores of 60 or above are generally considered clinically significant, and changes of 10 points or more (e.g., between pre-treatment and post-treatment) are considered clinically significant changes.
  units on a scale | 66.02 (14.85) | 72.98 (14.64) | 67.11 (17.83)
Posttraumatic Cognitions Inventory (PTCI) [Mean (Standard Deviation); unit: units on a scale] — The PTCI is a self-report questionnaire about thoughts following traumatic events. There are 33 scored items, each with response categories from 1 (Totally Disagree) to 7 (Totally Agree), summed to create the total score. Thus, the total score ranges from 7 to 231. Higher scores reflect higher levels of negative cognitions.
  units on a scale | 3.14 (1.07) | 3.78 (1.07) | 3.45 (1.13)
State-Trait Anxiety Inventory State Scale (STAI-S) [Mean (Standard Deviation); unit: units on a scale] — The STAI-S is a self-report questionnaire about state (present state) anxiety. There are 20 scored items, each with response categories from 1 (Not at All) to 4 (Very Much So). Some items (e.g., "I feel calm") are reversed scored so that the total score appropriately reflects state anxiety. Thus, the total score ranges from 20 to 80. Higher scores reflect higher levels of state anxiety.
  units on a scale | 44.46 (5.46) | 41.67 (6.13) | 43.08 (5.96)
Sheehan Disability Scale (SDS) [Mean (Standard Deviation); unit: units on a scale] — The SDS is a self-report questionnaire about functioning. There are 3 scored items (Work/School; Social Life; and Family Life/Home Responsibilities), each with response categories from 0 (zero; Not at All) to 10 (Extremely). Thus, the total score ranges from 0 to 30. Higher scores reflect lower (poorer) levels of functioning.
  units on a scale | 18.15 (8.03) | 18.83 (7.95) | 18.19 (8.09)
Global Neuropsychological Deficits (Standardized, Composite) [Mean (Standard Deviation); unit: standardized units on a scale] — Among our battery of seven neuropsychological tests, we worked with our neuropsychologist to choose 13 key scales. We used a conversion system to equally weight areas where there were large deficits, even if there were only one or two deficits, to prevent such scores from being minimized among the large range of T scores for the other scales. We converted T scores as follows: >40 = 0; 35-39 = 1; 30-34 = 2; 25-29 = 3; 20-24 = 4; < 20 = 5. Higher scores mean a higher global cognitive deficit.
  standardized units on a scale | .32 (.33) | .42 (.41) | .38 (.38)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Checklist (PCL)
Description: The PTSD Checklist is a self-report questionnaire about PTSD symptoms. The version used in this study is called the PCL-S, which denotes a specific traumatic event for subjects to respond to. There are 17 items, each with response categories from 1 to 5. Thus, the total score ranges from 17 to 85. Higher scores reflect higher levels of PTSD symptoms, and a score of 50 or above is commonly interpreted to designate clinically significant PTSD symptoms.
Time Frame: Pre-treatment, post-treatment, and 6-month follow-up
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT)
Number analyzed (Participants) | 41 | 46
units on a scale
  Baseline | 57.46 (12.66) | 59.98 (11.80)
  Post-Treatment | 47.00 (18.91) | 58.06 (12.31)
  6-Month Follow-Up | 58.37 (13.77) | 58.31 (10.88)

2. Secondary Outcome: Posttraumatic Cognitions Inventory (PTCI)
Description: The PTCI is a self-report questionnaire about thoughts following traumatic events. There are 33 scored items, each with response categories from 1 (Totally Disagree) to 7 (Totally Agree), summed to create the total score. Thus, the total score ranges from 7 to 231. Higher scores reflect higher levels of negative cognitions.
Time Frame: Pre-treatment, post-treatment, and 6-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT)
Number analyzed (Participants) | 41 | 46
units on a scale
  Baseline | 3.14 (1.07) | 3.78 (1.07)
  Post-Treatment | 2.80 (1.08) | 3.72 (1.04)
  6-Month Follow-Up | 3.44 (1.09) | 3.84 (1.11)

3. Secondary Outcome: State-Trait Anxiety Inventory State Scale (STAI-S)
Description: The STAI-S is a self-report questionnaire about state (present state) anxiety. There are 20 scored items, each with response categories from 1 (Not at All) to 4 (Very Much So). Some items (e.g., "I feel calm") are reversed scored so that the total score appropriately reflects state anxiety. Thus, the total score ranges from 20 to 80. Higher scores reflect higher levels of state anxiety.
Time Frame: Pre-treatment, post-treatment, and 6-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT)
Number analyzed (Participants) | 41 | 46
units on a scale
  Baseline | 44.46 (5.46) | 41.67 (6.13)
  Post-Treatment | 42.64 (5.81) | 43.75 (5.10)
  6-Month Follow-Up | 43.72 (5.96) | 42.63 (7.07)

4. Primary Outcome: Patient Health Questionnaire Depression Subscale (PHQ-9)
Description: The PHQ-9 is a self-report questionnaire about depressive symptoms. There are 9 scored items, each with response categories from 0 (zero) to 3. Thus, the total score ranges from 0 to 27. Higher scores reflect higher levels of depressive symptoms, with interpretation as follows:
  0 (zero) No depression 1-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression
Time Frame: Pre-treatment, post-treatment, and 6-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT)
Number analyzed (Participants) | 41 | 46
units on a scale
  Baseline | 12.13 (6.57) | 15.12 (5.17)
  Post-Treatment | 10.88 (7.67) | 14.80 (5.75)
  6-Month Follow-Up | 13.12 (6.15) | 13.92 (6.42)

5. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: The SDS is a self-report questionnaire about functioning. There are 3 scored items (Work/School; Social Life; and Family Life/Home Responsibilities), each with response categories from 0 (zero; Not at All) to 10 (Extremely). Thus, the total score ranges from 0 to 30. Higher scores reflect lower (poorer) levels of functioning.
Time Frame: Pre-treatment, post-treatment, and 6-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT)
Number analyzed (Participants) | 41 | 46
units on a scale
  Baseline | 18.15 (8.03) | 18.83 (7.95)
  Post-Treatment | 15.31 (8.89) | 18.77 (6.85)
  6-Month Follow-Up | 21.06 (7.44) | 17.71 (7.10)

6. Secondary Outcome: Global Neuropsychological Deficits (Standardized, Composite)
Description: Among our battery of seven neuropsychological tests, we worked with our neuropsychologist to choose 13 key scales. We used a conversion system to equally weight areas where there were large deficits, even if there were only one or two deficits, to prevent such scores from being minimized among the large range of T scores for the other scales. We converted T scores as follows: >40 = 0; 35-39 = 1; 30-34 = 2; 25-29 = 3; 20-24 = 4; < 20 = 5. Higher scores mean a higher global cognitive deficit.
Time Frame: Pre-treatment, post-treatment
Measure: Mean (Standard Deviation); unit: standardized units on a scale
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT)
Number analyzed (Participants) | 41 | 46
standardized units on a scale
  Baseline | .32 (.33) | .42 (.41)
  Post-Treatment | .35 (.42) | .40 (.42)

7. Primary Outcome: Clinician-Administered PTSD Scale Severity Score (CAPS)
Description: The CAPS is a clinician-administered interview about PTSD symptoms. There are 17 scored items for PTSD severity, each with response categories from 0 (zero) to 4 separately for both frequency and severity. Thus, each item can receive a score of 0 (zero) to 8, and the total severity score ranges from 0 to 136. Higher scores reflect higher levels of PTSD symptoms. Scores of 60 or above are generally considered clinically significant, and changes of 10 points or more (e.g., between pre-treatment and post-treatment) are considered clinically significant changes.
Time Frame: Pre-treatment, post-treatment, and 6-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT)
Number analyzed (Participants) | 41 | 46
units on a scale
  Baseline | 66.02 (14.85) | 72.98 (14.64)
  Post-Treatment | 48.48 (24.58) | 64.45 (15.32)
  6-Month Follow-Up | 29.16 (34.20) | 37.40 (32.74)

ADVERSE EVENTS:
Arm/Group | Prolonged Exposure Therapy (PE) | Relaxation Training (RT)
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/46
Other Adverse Events (participants affected / at risk) | 0/41 | 0/46

LIMITATIONS AND CAVEATS:
Early termination leading to smaller numbers of subjects analyzed at post-treatment and follow-up; Results generalize only to older male combat veterans who were treatment-seeking for PTSD

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No